CLINICAL TRIAL: NCT03673280
Title: Comparison Between Intrathecal Morphine and Quadratus Lumborum Block for Postpartum Analgesia of Elective Cesareans.
Brief Title: Quadratus Lumborum in Cesarean Section Trial
Acronym: QUALICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Hermann dos Santos Fernandes, MD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CAAE 90600818.0.0000.0068
Record Dates: First submitted 2018-09-03; First posted 2018-09-17 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Analgesia
Keywords: intrathecal morphine; quadratus lumborum block; cesarean c-section; postoperative pain; chronic pain
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Clinical, analytical, prospective, randomized trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Classical spinal anesthesia (Placebo Comparator): Patients allocated to this group will receive spinal anesthesia with bupivacaine 12.5mg, Fentanyl 20mcg and Morphine 80mcg + placebo quadratus lumborum block.
  Interventions: Procedure: Quadratus Lumborum Block
- Spinal anaesthesia with block (Experimental): Patients allocated to this group will receive spinal anesthesia with bupivacaine 12.5mg, Fentanyl 20mcg + quadratus lumborum block.
  Interventions: Procedure: Quadratus Lumborum Block
- Classical anaesthesia plus block (Experimental): Patients allocated to this group will receive spinal anesthesia with bupivacaine 12.5mg, Fentanyl 20mcg and Morphine 80mcg + quadratus lumborum block.
  Interventions: Procedure: Quadratus Lumborum Block

INTERVENTIONS:
Procedure: Quadratus Lumborum Block — Instead of using morphine in the classical spinal anaesthesia we will be performing in the experimental group the Quadratus Lumborum Block
  Other Names: Remove morphine from the spinal block

SUMMARY:
Postoperative pain of a caesarean section may be of high intensity, especially in the first 48 hours after the procedure, which affects the mother / newborn relationship, in addition to having the potential to progress to chronic pain. The use of intrathecal morphine is effective in post-caesarean analgesia, but carries unwanted side effects, including nausea, vomiting, urinary retention and pruritus. Therefore, alternative techniques of analgesia become necessary.

First described in 2007, ultrasound-guided quadratus lumborum (QL) block has gained prominence due to its analgesic superiority to the TAP block. Besides providing somatic analgesia, it also seems to inhibit visceral pain because the local anesthetic reaches the paravertebral space, this was observed by magnetic resonance imaging with contrast medium injected at the QL block site.

DETAILED DESCRIPTION:
C-section is one of the most performed surgical procedures in the world, and presents great potential for postoperative pain, especially in the first 48 hours. Pain in this period represents a risk for evolution to chronic pain, but its incidence is still very divergent when comparing the studies, ranging from 1% to 18%.

The use of intrathecal morphine (MIT) is consecrated as a first-choice method of analgesia for post-partum cesarean delivery; however, its use carries relevant side effects for the puerpera, such as pruritus, nausea, urinary retention and , more rarely, respiratory depression. In the last decade, new adjunctive forms of postoperative analgesia have become more popular, such as regional blockades, highlighting the blockage of the Transversus Abdominis plane block (TAP) and the Quadratus Lumborum block (QL), taking as benefits the prolonged analgesia they provide and the low incidence of side effects. Another factor that contributes to the popularization of regional blocks is the increasing availability of ultrasound devices in the anesthetic-surgical environment. Studies evaluating TAP block after cesarean section performed under spinal anesthesia have shown a discrete benefit in decreasing postoperative opioid consumption in addition to improving pain scores. When comparing MIT with TAP block, the superiority of MIT is due to visceral analgesia while TAP block is restricted to abdominal wall analgesia.

Ultrasound-guided Lumbar Quadrant blockade has gained prominence due to its analgesic superiority over the TAP block, because in addition to providing somatic analgesia it also seems to inhibit visceral pain since the local anesthetic reaches the paravertebral space, this was observed by magnetic resonance imaging with contrast injected at the site of the QL block.

Reviewing the literature in 2018, there are no clinical trials comparing the use of intrathecal morphine with the quadratus lumborum block.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Minimum gestational age of 37 weeks with a single fetus
* Patients scheduled for elective cesarean section through a Pfannenstiel incision under spinal anesthesia
* American Society of Anesthesiology physical status (ASA) II
* Body mass index (BMI) under 40 kg/m²
* No use of opioids for the past 4 weeks
* No history of psychotropic drug use
* No contraindication for any of the medications involved in the study
* No previously known malformations of the fetus
* No previous history of chronic pain

Exclusion Criteria:

* Difficulty in understanding how to use the patient-controlled analgesia (PCA) device
* Study protocol violation
* Patient decision to withdraw participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | 24 hours
  Evaluate pain in the postoperative period with to the consumption of morphine through PCA (patient controlled analgesia) pump.
Pain intensity | 24 hours
  Verbal numeric scale

SECONDARY OUTCOMES:
Nausea and Vomiting | 24 hours
  Evaluate the incidence of nausea and vomiting between the groups through referred nausea scale from none, mild, moderate or severe.
Pruritus | 24 hours
  Evaluate the incidence of pruritus between the groups through pruritus referred scale from none, mild, moderate or severe.
Chronic pain | 3 months
  Evaluate the incidence of chronic pain between the groups through patient referred presence or absence of pain.
Urinary retention | 24 hours
  Evaluate the incidence of urinary retention between the groups through patient referred presence or absence of urinary retention.

CONTACTS AND LOCATIONS:
Overall Officials: Hermann S Fernandes, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided